CLINICAL TRIAL: NCT02901288
Title: Shortened Regimens for First Diagnosed Smear Positive Drug Susceptible Pulmonary Tuberculosis: a Randomised Controlled Non-inferiority Trial
Brief Title: Shortened Regimens for Drug-susceptible Pulmonary Tuberculosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chest Hospital (Other)
Collaborators: Hubei Provincial Center for Disease Control and Prevention (Other); Centre for Tuberculosis Control of Guangdong Province (Unknown); Hunan Institute For Tuberculosis Control (Unknown); Anhui Chest Hospital (Other); Guangxi Zhuang Autonomous Region Center for Disease Prevention and Control (Other Government); Wuhan Institute for Tuberculosis Control (Other); Shanghai Pulmonary Hospital, Shanghai, China (Other); Shenyang Chest Hospital (Other); Changchun Infectious Disease Hospital (Unknown); First Affiliated Hospital of Xinjiang Medical University (Other); Public Health Clinical Center of Chengdu (Unknown); Taiyuan Fourth People's Hospital (Unknown); The Sixth People's Hospital of Nantong (Unknown); The Tuberculosis Prevention and Treatment Hospital of Shanxi Province (Unknown); Beijing Research Institute for Tuberculosis Control (Unknown); Infectious Disease Prevention Hospital in Heilongjiang Province (Unknown); The Third People's Hospital of Zhenjiang (Unknown); Tianjin centers for Disease Control and Prevention (Unknown); Harbin Chest Hospital (Unknown); Chest of Hospital of Xinjiang Uygur Autonomous Region of the PRC (Unknown); Heilongjiang Province center for tuberculosis Control and Prevention (Unknown); Tianjin Haihe Hospital (Other); The Infectious Disease Hospital of Wangkai Zaozhuang (Unknown); The Third People's Hospital of Kunming City (Unknown); Kaifeng Central Hospital (Other); The Infectious Hospital of Hebi (Unknown); Pulmonary Hospital of Lanzhou (Unknown); The Fourth People's Hospital of Ningxia Autonomous Region (Unknown); The Fourth People's Hospital of Qinghai Province (Other); The Fifth People's Hospital of Suzhou (Other); Chongqing Infectious Disease Medical Center (Unknown); Tuberculosis Hospital in Jilin Province (Unknown); Sixth People's Hospital of Nanyang City (Unknown); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Tang Shenjie, Director, TB Department, Beijing Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015ZX10003001
Record Dates: First submitted 2016-09-02; First posted 2016-09-15 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Tuberculosis, Pulmonary
Keywords: pulmonary tuberculosis; shortened regimen; clinical trial
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Isoniazid; Rifampin; Pyrazinamide; Ethambutol; Levofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- experimental group1 (Experimental): The experimental group1 all oral regimen is consisted of isoniazid,rifampin, pyrazinamide, ethambutol and levofloxacin for 4.5 months.
  Dosage: isoniazid 300mg(given once daily), rifampin 450mg(less than 50kg,given once daily)or 600mg(more than 50kg,given once daily), pyrazinamide 1500mg((less than 50kg,given once daily)or 30mg/kg(more than 50kg,once daily), ethambutol 750mg (less than 50kg,once daily) or 1000mg (more than 50kg,once daily), levofloxacin 600mg(less than 50kg,given once daily) or 800mg(more than 50kg,once daily).
  Interventions: Drug: Isoniazid; Drug: Rifampicin; Drug: Pyrazinamide; Drug: Ethambutol; Drug: Levofloxacin
- experimental group2 (Experimental): The experimental group2 all oral regimen consisted of isoniazid,rifampin, pyrazinamide, and ethambutol for 4.5 months. The dosage of isoniazid,rifampin, pyrazinamide, and ethambutol is as same as that of control regimen.
  Interventions: Drug: Isoniazid; Drug: Rifampicin; Drug: Pyrazinamide; Drug: Ethambutol
- Control regimen group (Active Comparator): The control all oral regimen consisted of isoniazid,rifampin, pyrazinamide, and ethambutol during the intensive phase of treatment (2 months), followed by isoniazid and rifampin during the continuation phase (4 months).
  Dosage: isoniazid 300mg(given once daily), rifampin 450mg(less than 50kg,given once daily)or 600mg(more than 50kg,given once daily), pyrazinamide 1500mg((less than 50kg,given once daily)or 30mg/kg(more than 50kg,once daily), ethambutol 750mg (less than 50kg,once daily) or 1000mg (more than 50kg,once daily).
  .
  Interventions: Drug: Isoniazid; Drug: Rifampicin; Drug: Pyrazinamide; Drug: Ethambutol

INTERVENTIONS:
Drug: Isoniazid — Isoniazid is a widely used anti-tuberculosis medication. Its primary action is to inhibit the synthesis of long-chain mycolic acids, which are unique components of mycobacterial cell wall.
Drug: Rifampicin — Rifampicin is a widely used anti-tuberculosis medication.
Drug: Pyrazinamide — Pyrazinamide is a commonly used medication for tuberculosis, with bactericidal effect against intracellular mycobacterium tuberculosis.
Drug: Ethambutol — Ethambutol is a widely used medicine in anti-TB regimens with bacteriostatic effect against M. tb.
Drug: Levofloxacin — Levofloxacin is a commonly used antimicrobial for TB and other infections, which acts on the DNA-DNA-gyrase complex and topoisomerase IV. It is the S (-) enantiomer of the racemic active substance ofloxacin.
  Other Names: Cravit
  Arms: experimental group1

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of two shortened regimens for newly diagnosed smear positive drug susceptible pulmonary tuberculosis in comparison to World Health Organization recommended standard 6-month regimen.

DETAILED DESCRIPTION:
1. Design: The study is a multi-center, randomized,controlled non-inferiority trial.
2. Population: patients with newly diagnosed drug-susceptible pulmonary TB who fulfill the inclusion and exclusion criteria.
3. Investigational regimens:

   Experimental group 1 regimen consists of levofloxacin, isoniazid , rifampicin,ethambutol and pyrazinamide for 4.5 months.

   Experimental group 2 regimen consists of isoniazid, rifampicin, ethambutol and pyrazinamide for 4.5 months.

   The control group is WHO recommended regimen conmposed of isoniazid , rifampicin, ethambutol and pyrazinamide for 2 months, followed by isoniazid , rifampicin for 4 months.

   Dosage: isoniazid 300mg(given once daily), rifampin 450mg(less than 50kg,given once daily)or 600mg(more than 50kg,given once daily), pyrazinamide 1500mg(less than 50kg,given once daily)or 30mg/kg(more than 50kg,once daily), ethambutol 750mg (less than 50kg,once daily) or 1000mg (more than 50kg,once daily), levofloxacin 600mg(less than 50kg,given once daily) or 800mg(more than 50kg,once daily)..
4. Trial objectives: to evaluate that shortened regimens is not inferior to standard treatment in terms of efficacy and safety for new smear positive pulmonary TB patients.
5. Primary and Secondary outcome measures:

   The primary efficacy outcome measures include (a)the percentage of participants with TB recurrence/relapse by 24 months after the end of treatment;(b) percentage of participants with treatment failure at either 4.5 months or 6 months after randomization. (a) Time to sputum smear or culture conversion within intensive phase.(b) Sputum smear conversion proportion at the treatment completion. (c) Number of adverse drug reaction occurring during treatment or follow-up period. (d) Radiological manifestation change of TB lesion or cavity.(e) Patients adherence rate.
6. Sample Size:

   Approximately 3900 participants will be enrolled and randomized with 1:1:1 ratio into either Experimental group1, Experimental group2 or control group.
7. Blinding:

   The study is an open-label study.
8. Assessment and follow-up:

All patients will be followed by to 2 years after completion of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Is willing and able to give informed consent to participate in the trial treatment and follow-up (signed or witnessed consent if the patient is illiterate).
2. Is aged 18-65 years.
3. Has twice positive acid-fast bacilli(AFB) sputum smear or positive sputum culture result, along with chest x-ray imaging consistent with active pulmonary tuberculosis.
4. Newly diagnosed cases receiving anti-TB treatment for less than one month
5. Urine Human Chorionic Gonadotropin(U-HCG) negative and must agree to use effective contraception during the trial period.
6. Has Alanine aminotransferase（ALT）and Total bilirubin（TBil） less than 2 times the upper limit of normal ; has Creatinine clearance rate （CrCI） more than 30ml/min; has Hemoglobin more than 7.0g/dL; has Platelet（PLT）more than 50 x10^9/L before study entry.

Exclusion Criteria:

1. Concomitant severe cardiovascular, liver, kidney, nervous system, hematopoietic system and other diseases, or concomitant neoplastic diseases. Or extensive lesion with respiratory insufficiency.
2. Uncontrolled diabetes mellitus.
3. Concomitant mental disorders.
4. Is HIV positive.
5. Is critically ill, and in the judgment of the investigator, not fit for the study or unlikely to complete the full course of study.
6. Is known to be pregnant or breast-feeding.
7. Is unable or unwilling to comply with the treatment, assessment, or follow-up schedule.
8. Is taking any medications contraindicated with the medicines in any trial regimen of the study.
9. Has a known allergy to any drug of treatment regimens.
10. Is currently taking part in another trial.
11. Has a QTc interval more than 480ms.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3900 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The percentage of participants with TB recurrence/relapse by 24 months after the end of treatment. | 24 months after treatment completion for all 3 groups
Percentage of participants with treatment failure at either 4.5 months or 6 months after randomization. | 4.5 months after randomization for experimental group1 and 2; 6 months after randomization for control group

SECONDARY OUTCOMES:
Treatment adverse reactions occuring | An average of 6 months for control group and 4.5 months for experimental group1 and 2 during treatment and 24 months after treatment completion.
Time to sputum smear or culture conversion within intensive phase . | An avergae of 2-3 months after randomization.
Sputum smear or culture conversion proportion at the treatment completion. | An average of 6 months for control group while 4.5 months for experimental group 1 and 2.
Radiological manifestation change of TB lesion or cavity. | An average of 6 months during treatment and 24 months after treatment completion.
Patiens adherence rate | An average of 6 months during treatment and 24 months after treatment completion.

CONTACTS AND LOCATIONS:
Overall Officials: Shenjie Tang, MD, Principal Investigator — Beijing Chest Hospital
Locations (35):
- China (35):
  - Anhui Chest Hospital, Hefei, Anhui
  - Beijing Research Institute for Tuberculosis Control, Beijing, Beijing Municipality
  - Beijing Chest Hospital,Capital Meical University, Beijing, Beijing Municipality
  - Chongqing Infectious Disease Medical Center, Chongqing, Chongqing Municipality
  - Pulmonary Hospital of Lanzhou, Lanzhou, Gansu
  - Centre for Tuberculosis Control of Guangdong Province, Guangzhou, Guangdong
  - Guangxi Center for Disease Prevention and Control, Nanning, Guangxi
  - HeBei Province Center for Disease Prevention and Control, Shijiazhuang, Hebei
  - Heilongjiang Province center for tuberculosis Control and Prevention, Haerbin, Heilongjiang
  - Harbin Chest Hospital, Harbin, Heilongjiang
  - Infectious Disease Prevention Hospital in Heilongjiang Province, Harbin, Heilongjiang
  - The Infectious Hospital of Hebi, Hebi, Henan
  - Kaifeng Pulmonary Disease Hospital, Kaifeng, Henan
  - Sixth People's Hospital of Nanyang City, Nanyang, Henan
  - The First Affiliated Hospital of Xinxiang Medical University, Xianxiang, Henan
  - Wuhan medical treatment center, Wuhan, Hubei
  - Wuhan Institute For Tuberculosis Control, Wuhan, Hubei
  - Hunan Institute For Tuberculosis Control, Changsha, Hunan
  - The Sixth People's Hospital of Nantong, Nantong, Jiangsu
  - The Fifth People's Hospital of Suzhou, Suzhou, Jiangsu
  - The Third People's Hospital of Zenjiang, Zhenjiang, Jiangsu
  - Changchun Infectious Disease Hospital, Changchun, Jilin
  - Tuberculosis Hospital in Jilin Province, Jilin, Jilin
  - China Shenyang Chest Hospital, Shenyang, Jilin
  - The Fourth People's Hospital of Ningxia Autonomous Region, Yinchuan, Ningxia
  - The 4th People's Hospital of Qinghai Province, Xining, Qinghai
  - The Infectious Disease Hospital of Wangkai Zaozhuang, Tengzhou, Shandong
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Taiyuan Fourth People's Hospital, Taiyuan, Shanxi
  - The Tuberculosis Prevention and Treatment Hospital of Shanxi Province, Xi’an, Shanxi
  - Public Health Clinical Center of Chengdu, Chengdu, Sichuan
  - Tianjin Haihe Hospital, Tianjin, Tianjin Municipality
  - Tianjin centers for Disease Control and Prevention, Tianjin, Tianjin Municipality
  - Chest of Hospital of Xinjiang Uygur Autonomous Region of the PRC, Ürümqi, Xinjiang
  - The Third People's Hospital of Kunming City, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao M, Gao J, Du J, Liu Y, Zhang Y, Ma L, Mi F, Li L, Tang S; Trial Team. Efficacy of ultra-short course chemotherapy for new smear positive drug susceptible pulmonary tuberculosis: study protocol of a multicenter randomized controlled clinical trial. BMC Infect Dis. 2017 Jun 19;17(1):435. doi: 10.1186/s12879-017-2505-7. PMID 28629333
- [Derived] Pease C, Hutton B, Yazdi F, Wolfe D, Hamel C, Quach P, Skidmore B, Moher D, Alvarez GG. Efficacy and completion rates of rifapentine and isoniazid (3HP) compared to other treatment regimens for latent tuberculosis infection: a systematic review with network meta-analyses. BMC Infect Dis. 2017 Apr 11;17(1):265. doi: 10.1186/s12879-017-2377-x. PMID 28399802